CLINICAL TRIAL: NCT03509935
Title: Use of Bedside Ultrasonography on the Incidence of Acute Renal Failure in High-risk Surgical Patients: Randomized Clinical Trial
Brief Title: Use of Bedside Ultrasonography on the Incidence of Acute Renal Failure in High-risk Surgical Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Minas Gerais (Other)
Responsible Party: Principal Investigator, Vandack Alencar Nobre, Principal Investigator, Federal University of Minas Gerais
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: US to guide ressuscitation
Record Dates: First submitted 2018-04-12; First posted 2018-04-27 (Actual); Last update posted 2020-07-22 (Actual); Status verified 2018-04

CONDITIONS: Acute Kidney Injury
Keywords: ultrasound,; high-risk surgery; intensive care
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Ultrasound Group (Experimental): Patients will be submitted to Ultrasound protocol, namely:
  1. In the first 6 to 12 hours of admission to ICU
  2. Second US after 12-24 hours of inclusion.
  3. Third US after 24-48 hours of inclusion.
  Protocol:
  * US 4 pulmonary quadrants in each hemithorax: anterior and lateral, upper and lower regions.
  * US inferior vena cava, collapsability or distensibility index according to the patient's conditions, in spontaneous or controlled ventilation, respectively.
  * Cardiac US: subjective evaluation of contractility between normal, reduced or severely reduced.
  The US findings will be communicated to the attending physicians who will conduct the patient, according to the protocol, recommending the administration of volume or not, and the use of vasopressors and/or inotropic drugs.
  Interventions: Other: Intervention Ultrasound Group
- Control Group (No Intervention): Patients randomized to this group will receive care according to the indication of the attending physicians, composed mainly of intensive care physicians, without bedside US. Patients may be submitted to echocardiographic, abdominal and vascular examinations, among others, requested to ultrasound service, according to the indication.

INTERVENTIONS:
Other: Intervention Ultrasound Group — Protocol:
  * US 4 pulmonary quadrants in each hemithorax: anterior and lateral, upper and lower regions (figure 1)
  * US inferior vena cava, collaborative index or distensibility according to the patient's conditions, in spontaneous or controlled ventilation, respectively.
  * Cardiac US: subjective evaluation of contractility in normal, discreetly reduced or severely reduced.
  Arms: Intervention Ultrasound Group

SUMMARY:
The mortality and postoperative complications of high risk surgeries vary in the different series. The management of this group of patients in intensive care unit (ICU) is fundamental to improve these outcomes. The objective of this study will be to evaluate whether the use of bedside ultrasound has an impact on the management of this group of patients with a consequent reduction in the incidence of acute renal failure in ICU and, secondarily, the incidence of associated complications. All adult patients (≥ 18 years old) admitted to ICU at Hospital das Clinicas of UFMG in the immediate postoperative period of major surgery with indication of ICU monitoring will be included and randomly randomized to the control or intervention group. The control group will be conducted by the intensive care physicians in charge without the US, while the second group will be conducted based in US findings. The US protocol will consist of a pulmonary US in four windows in each hemithorax , qualitative assessment of contractility and variation of inferior vena cava diameter. The primary outcome will be the development of acute renal failure as measured by the KDIGO score. Secondary outcomes will be length of ICU and hospital stay, ICU and 28 days mortality, length spent in mechanical ventilation, accumulated water balance, noradrenaline and dobutamine dose. Serum and urinary biomarkers will also be evaluated. Key words: ultrasound, high-risk surgery, intensive care

DETAILED DESCRIPTION:
This is a single-center randomized clinical trial to be performed at the Adult Intensive Care Unit (ICU) of the Clinical Hospital of the Federal University of Minas Gerais, Belo Horizonte. The ICU is a clinical-surgical unit that has 18 beds with admission of approximately 100 patients per month, being 70% surgical patients and 30% clinical patients. Postoperative patients who meet the inclusion criteria reported below will be randomized to guide therapy according to ultrasound findings at the bedside versus a group that will not perform this method. Serum and urine samples will be collected in three times: admission (T0), after 12 hours (T1) and after 24 hours (T2) to analysed urine and serum biomarkers.

ELIGIBILITY:
Inclusion Criteria:

* Age equal or superior to 18 years.
* Major surgeries requiring ICU admission associated with one of the following criteria:

  * Use of vasoactive drugs
  * Use of inotropic drugs
  * Mean blood pressure less than 65 mmHg or SBP <90 mmHg.
  * Hyperlactatemia> 2 mmol / L
  * Heart rate> 90 bpm.
  * Invasive mechanical ventilation required for at least 6 hours at the time of inclusion.
  * Hypoxia: satO2 <92% in ambient air.
  * Length of surgery greater than 4 hours.
  * Request for transfusion of blood products in a surgical block
  * Oliguria during procedure, defined as diuresis <0.5 ml/kg/h.

Exclusion Criteria:

Patients who do not agree to the terms of the

* Dying patients with impending death in the first 24 hours
* Patients in a previous renal replacement therapy program

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 111 (Actual)
Dates: Start 2018-03-12 (Actual); Primary Completion 2019-03-31 (Actual); Study Completion 2019-03-31 (Actual)

PRIMARY OUTCOMES:
Acute renal failure (ARF) | One week
  Creatinine elevation or oliguria according to KDIGO classification Impact in the incidence of ARF in major surgeries

SECONDARY OUTCOMES:
Volume replacement within the first 36 hours. | 36 hours
  Quantity of volume administered during first 36 hours of admission in ICU
Use of vasopressor drugs. | 36 hours
  vasopressor drugs requirement mcg/kg/min
Use of inotropic drugs. | 36hours
  Inotropic drug requirement in mcg/kg/min
Length of invasive mechanical ventilation | 36 hours
  Days spent in invasive mechanical ventilation
Length of ICU stay | 28 days
  Days spent in ICU
Length of Hospital stay | 28 days
  Days spent in Hospital
Mortality in ICU | 28 days
  Any cause of mortality during ICU stay
28 days mortality | 28 days
  Any cause of mortality in 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Vandack Nobre, PhD, Principal Investigator — Hospital das Clincias UFMG
Locations (1):
- Hospital das Clínicas - Universidade Federal de Minas Gerais, Belo Horizonte, Minas Gerais, Brazil

IPD SHARING:
Plan to Share IPD: No